CLINICAL TRIAL: NCT06861140
Title: Untersuchung Des Einflusses Einer Tryptophanreichen Diät Auf Das Therapeutische Potential Von Probiotika Nach Antibiotischer Therapie Bei Chronischer Pouchitis (Try Pro Pouch). Eine Prospektive Randomisierte Kontrollierte Doppelblinde Interventionsstudie
Brief Title: Exploring the Influence of Trptophan on the Treatment of Pouchitis
Acronym: TryProPouch
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-101427-BO-ff; Intramural funding (Other Grant/Funding Number: I. Medizinische Klinik und Poliklinik, UKE)
Record Dates: First submitted 2025-02-23; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Pouchitis
Keywords: Pouchitis; Antibiotics; Probiotics; Tryptophan; Metabolites
MeSH Terms: conditions — Pouchitis | interventions — Tryptophan

STUDY DESIGN:
Intervention Model Description: Interventional, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: care providers, Investigators and Outcome Assessors are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): regular treatment of pouchitis with consecutive application of antibiotics and probiotics, followed by placebo.
  Interventions: Other: Placebo
- Intervention (Experimental): regular treatment of pouchitis with consecutive application of antibiotics and probiotics, additional supplementation of tryptophan (25mg/kg bodyweight)
  Interventions: Dietary Supplement: Tryptophan 25mg/kg bodyweight

INTERVENTIONS:
Dietary Supplement: Tryptophan 25mg/kg bodyweight — Tryptophan is supplemented during the treatment of chronic pouchitis with pro- and antibiotics
  Arms: Intervention
Other: Placebo — standard treatment of chronic pouchitis using pro- and antibiotics.
  Arms: Placebo

SUMMARY:
Patients with a pouch frequently suffer from chronic inflammation of the intestinal tract, called pouchitis. Pouchitis is routienly treated with repeated courses of antibiotics and probiotics, which does not stop the inflammation from recurring and exposes the patients to the risk of developing antibiotic -resistant pouchitis. Experimental data suggest that the effectiveness of the antibiotic and probiotic treatment can be prolonged by high consumption of trypotophan, an aminoacid present in everyday food. The Try Pro Pouch study aims to compare the consumption of high amounts of tryptophan against placebo in patients with pouchitis.

DETAILED DESCRIPTION:
Participants with chronic pouchitis receive either a weight adapted supplement containing etiher trypotophan or a placebo after completing the standard treatment with antibiotics or probiotics for their pouchitis. Endoskopy will be performed, stool and blood will be sampled, symptoms will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Pouchitis (PDAI >= 7)
* indication for the application of antibiotics and probiotics
* Age >=18 years
* Informed consent

Exclusion Criteria:

* major surgery planned druing the intervention
* high risk for malnutrition (NRS 2002 >=3/ BMI <18,5 kg/m^2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Increase of the proportion of FoxP3+ CD4+ T cells in gut biopsies | from enrollent to end of treatment at 12 weeks
  Biopsies of individuals receiving tryptophan or placebot will be analysed by Flow-Cytometry or sequencing. We aim to detect an lasting increase of the proportion of FoxP3+ CD4+ T cells in the mucosa of individuals receiving tryptophan, but not in those receiving placebo.

SECONDARY OUTCOMES:
Increase of the frequency of Lactobacilli and Bifidobacilli in the gut microbiota | from enrollent to end of treatment at 12 weeks
  The microbiota composition will be analysed by 16sRNA sequencing. We aim to detect a relative increase of lactobacilli and bifidobacilli in all study participants following the consecutive treatment with anti- and probiotics.
Increase of 3-IPA-levels in blood and stool | from enrollent to end of treatment at 12 weeks
  3-IPA will be measured by ELISA in in the blood and stool of participants receiving tryptophan or placebo. We expect greater increase of systemic 3-IPA in individuals receiving tryptophan.
Higher rates of therapeutic response defined by PDAI | from enrollent to end of treatment at 12 weeks
  Endoscopy is performed before and after the intervention. We aim to reach better treatment response defined by lower PDAI, a histologic score of Pouchitis severity.
Decreased number of prescribed antibiotics druing follow-up | from enrollent to end of observation at 52 weeks
  The number of relapses, defined as repeated indication for antibiotics, during the observational follow-up will be counted. We aim to archive reduced number of antibiotic prescriptions indicated because of pouchitis in the intervention group during the one year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Huber, Prof. Dr. med., Principal Investigator — Universitätsklinkum Hamburg-Eppendorf, I. Medizinische Klinik und Poliklinik

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared without resonable request. If, after publication, researches ask for IPD for further analysis, anonymized data will shared.